CLINICAL TRIAL: NCT05643235
Title: Implanted Loop Recorders (ILR) for the Detection and Management of Arrhythmia in Patients Treated With Bruton Tyrosine Kinase (BTK) Inhibitors
Brief Title: Implanted Loop Recorders for Detection and Management of Arrhythmia With Bruton Tyrosine Kinase Inhibitors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Robert Copeland-Halperin, MD FACC, Assistant Professor of Cardiology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 22-0256; ERP-2021-12882 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Supraventricular Arrhythmia; Ventricular Arrhythmias and Cardiac Arrest; Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Keywords: Bruton tyrosine kinase (BTK); Chronic Lymphocytic Leukemia (CLL); Mantle Cell Lymphoma; Waldenstrom's macroglobulinemia; atrial fibrillation (AF); ventricular arrhythmia (VA); sudden cardiac death; ibrutinib; acalabrutinib; zanubrutinib; pirtobrutinib; Implanted Loop Recorder/Implanted Cardiac Monitor (ILR)
MeSH Terms: conditions — Atrial Fibrillation; Heart Arrest; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Single arm, prospective study of implanted loop recorders (ILR) for the detection of arrhythmia in patients initiating treatment with BTK inhibitors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients initiated on Bruton tyrosine kinase inhibitors, consenting to installment of ILR (Other): Patients free of documented arrhythmia initiating treatment with a BTK inhibitor who consent to monitoring using the Medtronic LINQ-2 implanted cardiac monitoring device (ILR) prior to initiating BTK inhibitor therapy.
  Interventions: Device: Medtronic LINQ-2 Insertable Cardiac Monitor (ILR)

INTERVENTIONS:
Device: Medtronic LINQ-2 Insertable Cardiac Monitor (ILR) — Patients initiating BTK inhibitors will be offered the option of monitoring using the Medtronic Insertable Cardiac Monitor (ILR). The device will be implanted by a certified and credentialed electrophysiologist to enable monitoring to begin at least 24 hours prior to the first administration of the BTK inhibitor. Monitoring data will be collected prospectively until the patient withdraws consent, the device is removed, or up to 60 months

SUMMARY:
This study will enroll patients initiating Bruton Tyrosine Kinase (BTK) inhibitors without history of documented arrhythmia while on therapy using the Medtronic LINQ-2 insertable cardiac monitor (ILR). The incidence of new onset atrial fibrillation (AF) and other arrhythmia will be determined. Actions taken in response to device detected arrhythmia will be recorded.

DETAILED DESCRIPTION:
This single arm, prospective non-blinded study will enroll 50 patients initiating treatment with BTK inhibitors (ibrutinib, acalabrutinib, zanubrutinib or pirtobrutinib) without documented arrhythmia prior to starting BTK inhibitor therapy, without contraindications to an implanted loop recorder (ILR). They will be offered the option of monitoring arrhythmias using the Medtronic LINQ-2 insertable cardiac monitor (ILR). Monitoring data will be collected prospectively until the patient withdraws consent, the device is removed, or up to 60 months. Investigators hope to obtain information on arrhythmia incidence including AF, ventricular arrhythmia (VA), and actions taken in response to awareness of such episodes.

ELIGIBILITY:
Inclusion Criteria:

* >18yo
* Willing to sign and date consent form,
* Willing to be remotely monitored
* Initiating BTK inhibitor for approved condition (i.e. CLL, Waldenstrom's, etc)
* Willing to have Medtronic cardiac monitor inserted to allow at minimum 24 hours continuous monitoring prior to initiating BTK inhibitor

Exclusion Criteria:

* Documented AF/VA in past 12 months
* Cerebral Vascular Accident (CVA) or Transient Ischemic Attack (TIA) in past year
* Has current implanted pulse generator, defibrillator, pacemaker, or resynchronization device
* heart surgery within past 90 days
* Myocardial Infarction within past 90 days
* Patient is taking an anti-arrhythmic or anticoagulant
* has concomitant condition that precludes safe participation in study (substance abuse, etc)
* Enrollment in separate study that could confound results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of device detected atrial fibrillation (AF) | at 18 months after start of BTK inhibitor
  Incidence of AF lasting 6 or more minutes at 18 months: each arrhythmic episode detected by the patient's device will be reviewed to determine if it is 1) an actual AF episode, and 2) is at least 6 minutes in duration.
Long term Incidence of device detected AF | up to 60 months after device implantation
  Incidence of AF lasting 6 or more minutes up to 60 months: each arrhythmic episode detected by the patient's device will be reviewed to determine if it is 1) an actual AF episode, and 2) is at least 6 minutes in duration.

SECONDARY OUTCOMES:
Incidence of device detected ventricular arrhythmia (VA) | at 18 months after start of BTK inhibitor
  Incidence of VA is defined as follows: greater than or equal to 3 sequential wide complex beats arising from the ventricles, rate > 100 beats per minute at 18 months after start of BTK inhibitor therapy.
BTK dose reduction or discontinuation due to device detected arrhythmia, assessed by chart review. | up to 60 months after device implantation
  Clinical actions including BTK dose reduction, interruption, discontinuation, or change in oncologic treatment by treating oncologist because of device detected arrhythmia.
Initiation of anticoagulation for AF detected by device monitoring, assessed by chart review | up to 60 months after device implantation
  Prescription of an approved anticoagulant drug (apixaban, dabigatran, rivaroxaban, edoxaban, warfarin, aspirin) for prevention of stroke/systemic embolism based on AF detected by ILR
Long term incidence of device detected ventricular arrhythmia (VA) | up to 60 months after device implantation
  Incidence of VA is defined as follows: greater than or equal to 3 sequential wide complex beats arising from the ventricles, rate > 100 beats per minute up to 60 months after device implant.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Copeland-Halperin, MD, Principal Investigator — Northwell Health; Haisam Ismail, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell (Northshore University/Long Island Jewish Hospitals), New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganatra S, Sharma A, Shah S, Chaudhry GM, Martin DT, Neilan TG, Mahmood SS, Barac A, Groarke JD, Hayek SS, Dani S, Venesy D, Patten R, Nohria A. Ibrutinib-Associated Atrial Fibrillation. JACC Clin Electrophysiol. 2018 Dec;4(12):1491-1500. doi: 10.1016/j.jacep.2018.06.004. Epub 2018 Aug 29. PMID 30573111
- [Background] Baptiste F, Cautela J, Ancedy Y, Resseguier N, Aurran T, Farnault L, Escudier M, Ammar C, Gaubert M, Dolladille C, Barraud J, Peyrol M, Cohen A, Paganelli F, Alexandre J, Ederhy S, Thuny F. High incidence of atrial fibrillation in patients treated with ibrutinib. Open Heart. 2019 May 8;6(1):e001049. doi: 10.1136/openhrt-2019-001049. eCollection 2019. PMID 31168393
- [Background] Guha A, Derbala MH, Zhao Q, Wiczer TE, Woyach JA, Byrd JC, Awan FT, Addison D. Ventricular Arrhythmias Following Ibrutinib Initiation for Lymphoid Malignancies. J Am Coll Cardiol. 2018 Aug 7;72(6):697-698. doi: 10.1016/j.jacc.2018.06.002. No abstract available. PMID 30072003
- [Background] Lampson BL, Yu L, Glynn RJ, Barrientos JC, Jacobsen ED, Banerji V, Jones JA, Walewska R, Savage KJ, Michaud GF, Moslehi JJ, Brown JR. Ventricular arrhythmias and sudden death in patients taking ibrutinib. Blood. 2017 May 4;129(18):2581-2584. doi: 10.1182/blood-2016-10-742437. Epub 2017 Feb 21. No abstract available. PMID 28223277
- [Background] Byrd JC, Hillmen P, O'Brien S, Barrientos JC, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Barr PM, Furman RR, Kipps TJ, Thornton P, Moreno C, Montillo M, Pagel JM, Burger JA, Woyach JA, Dai S, Vezan R, James DF, Brown JR. Long-term follow-up of the RESONATE phase 3 trial of ibrutinib vs ofatumumab. Blood. 2019 May 9;133(19):2031-2042. doi: 10.1182/blood-2018-08-870238. Epub 2019 Mar 6. PMID 30842083
- [Background] Tam CS, Opat S, D'Sa S, Jurczak W, Lee HP, Cull G, Owen RG, Marlton P, Wahlin BE, Sanz RG, McCarthy H, Mulligan S, Tedeschi A, Castillo JJ, Czyz J, Fernandez de Larrea C, Belada D, Libby E, Matous JV, Motta M, Siddiqi T, Tani M, Trneny M, Minnema MC, Buske C, Leblond V, Trotman J, Chan WY, Schneider J, Ro S, Cohen A, Huang J, Dimopoulos M. A randomized phase 3 trial of zanubrutinib vs ibrutinib in symptomatic Waldenstrom macroglobulinemia: the ASPEN study. Blood. 2020 Oct 29;136(18):2038-2050. doi: 10.1182/blood.2020006844. PMID 32731259
- [Background] Janssen Biotech I. Imbruciva Prescribing Information. Janssen Biotech, Inc. 2020. Accessed December 21, 2021. https://www.imbruvica.com/files/prescribing-information.pdf
- [Background] CALQUENCE PRESCRIBING INFORMATION (AstraZeneca Pharmaceuticals LP) (2019).
- [Background] Ltd BU. Brukinsa Prescribing Information. 2021.
- [Background] Munir T, Brown JR, O'Brien S, Barrientos JC, Barr PM, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Kipps TJ, Moreno C, Montillo M, Burger JA, Byrd JC, Hillmen P, Dai S, Szoke A, Dean JP, Woyach JA. Final analysis from RESONATE: Up to six years of follow-up on ibrutinib in patients with previously treated chronic lymphocytic leukemia or small lymphocytic lymphoma. Am J Hematol. 2019 Dec;94(12):1353-1363. doi: 10.1002/ajh.25638. Epub 2019 Oct 13. PMID 31512258
- [Background] Byrd JC, Hillmen P, Ghia P, Kater AP, Chanan-Khan A, Furman RR, O'Brien S, Yenerel MN, Illes A, Kay N, Garcia-Marco JA, Mato A, Pinilla-Ibarz J, Seymour JF, Lepretre S, Stilgenbauer S, Robak T, Rothbaum W, Izumi R, Hamdy A, Patel P, Higgins K, Sohoni S, Jurczak W. Acalabrutinib Versus Ibrutinib in Previously Treated Chronic Lymphocytic Leukemia: Results of the First Randomized Phase III Trial. J Clin Oncol. 2021 Nov 1;39(31):3441-3452. doi: 10.1200/JCO.21.01210. Epub 2021 Jul 26. PMID 34310172
- [Background] Medtronic. LINQ II LNQ22 ICM Clinician Manual. M974764A001D.
- [Background] Sakhi R, Theuns DAMJ, Szili-Torok T, Yap SC. Insertable cardiac monitors: current indications and devices. Expert Rev Med Devices. 2019 Jan;16(1):45-55. doi: 10.1080/17434440.2018.1557046. Epub 2018 Dec 11. PMID 30522350
- [Background] Sakhi R, Huurman R, Theuns DAMJ, Schinkel AFL, Assaf A, Szili-Torok T, Roos-Hesselink JW, Michels M, Yap SC. Incremental Value of an Insertable Cardiac Monitor in Patients with Hypertrophic Cardiomyopathy with Low or Intermediate Risk for Sudden Cardiac Death. Cardiology. 2021;146(2):207-212. doi: 10.1159/000512656. Epub 2021 Jan 21. PMID 33477163
- [Background] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Wachter R, Pouliot E, Ziegler PD; REVEAL AF Investigators. Incidence of Previously Undiagnosed Atrial Fibrillation Using Insertable Cardiac Monitors in a High-Risk Population: The REVEAL AF Study. JAMA Cardiol. 2017 Oct 1;2(10):1120-1127. doi: 10.1001/jamacardio.2017.3180. PMID 28842973
- [Background] Bernstein RA, Kamel H, Granger CB, Piccini JP, Sethi PP, Katz JM, Vives CA, Ziegler PD, Franco NC, Schwamm LH; STROKE-AF Investigators. Effect of Long-term Continuous Cardiac Monitoring vs Usual Care on Detection of Atrial Fibrillation in Patients With Stroke Attributed to Large- or Small-Vessel Disease: The STROKE-AF Randomized Clinical Trial. JAMA. 2021 Jun 1;325(21):2169-2177. doi: 10.1001/jama.2021.6470. PMID 34061145
- [Background] Sirichand S, Killu AM, Padmanabhan D, Hodge DO, Chamberlain AM, Brady PA, Kapa S, Noseworthy PA, Packer DL, Munger TM, Gersh BJ, McLeod CJ, Shen WK, Cha YM, Asirvatham SJ, Friedman PA, Mulpuru SK. Incidence of Idiopathic Ventricular Arrhythmias: A Population-Based Study. Circ Arrhythm Electrophysiol. 2017 Feb;10(2):e004662. doi: 10.1161/CIRCEP.116.004662. PMID 28183845